CLINICAL TRIAL: NCT07004374
Title: Comparative Effects of Instrument-Assisted Soft Tissue Mobilization and Percussion Vibration Therapy on Balance, Explosive Strength, and Functional Performance in Competitive Adolescent Rowers: A Randomized Controlled Trial
Brief Title: Effects of Soft Tissue Mobilization and Vibration Therapy in Competitive Rowers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Emre DANSUK, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-2942
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Balanced; Soft Tissue Injuries
Keywords: Rowing; Instrument-assisted soft tissue mobilization (IASTM); Percussion massage therapy; Balance; Explosive strength; Functional performance
MeSH Terms: conditions — Soft Tissue Injuries

STUDY DESIGN:
Intervention Model Description: This study is designed as a randomized controlled trial (RCT) with a parallel-group design to evaluate the comparative effects of two different therapeutic interventions-instrument-assisted soft tissue mobilization (IASTM) and percussion vibration therapy-on balance, explosive strength, and functional performance in adolescent competitive rowers.
  A total of 45 participants will be randomly assigned to one of three groups:
  Group 1: Vibration Therapy Group (percussion massage therapy at 33 Hz) Group 2: Soft Tissue Mobilization Group (Graston technique/IASTM) Group 3: Control Group (no intervention)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Participants in this group will not receive any intervention.
- Vibration Therapy (33 Hz) Group (Experimental): Participants receive percussion massage therapy (33 Hz) applied to the quadriceps and gastrocnemius muscles using a handheld massage device for 5 minutes per muscle group.
  Interventions: Device: a percussion massage gun
- Soft Tissue Mobilization Group (Experimental): Participants receive instrument-assisted soft tissue mobilization (IASTM, Graston technique) applied to the quadriceps and gastrocnemius muscles using stainless steel tools with standardized techniques (Sweep, Fan, Brush) for 6 minutes.
  Interventions: Device: specially designed stainless-steel instruments

INTERVENTIONS:
Device: a percussion massage gun — Participants receive percussion massage therapy (33 Hz) applied to the quadriceps and gastrocnemius muscles using a handheld massage device for 5 minutes per muscle group.
  Arms: Vibration Therapy (33 Hz) Group
Device: specially designed stainless-steel instruments — Participants receive instrument-assisted soft tissue mobilization (IASTM, Graston technique) applied to the quadriceps and gastrocnemius muscles using stainless steel tools with standardized techniques (Sweep, Fan, Brush) for 6 minutes.
  Arms: Soft Tissue Mobilization Group

SUMMARY:
This randomized controlled study aims to investigate the effects of instrument-assisted soft tissue mobilization (IASTM) and percussion massage therapy on balance, explosive strength, and functional performance in competitive adolescent rowers. A total of 45 participants aged 13-18 will be randomly assigned to one of three groups: vibration therapy group, soft tissue mobilization group, and control group. Interventions will target the quadriceps and gastrocnemius muscles. Outcome measures include the Y Balance Test, vertical jump, hop tests, and isometric muscle strength via myometry. The results of this study are expected to provide evidence-based insights into optimizing performance and injury prevention strategies in rowing athletes.

DETAILED DESCRIPTION:
Rowing is a high-performance sport that demands coordinated action of the upper and lower extremities, trunk muscles, and cardiovascular system. Due to repetitive pulling movements, rowers are prone to musculoskeletal overload injuries, particularly in the lower back, shoulders, knees, and ankles. Effective balance control and lower extremity explosive strength are critical for performance enhancement and injury prevention in rowing athletes. Soft tissue mobilization techniques and vibration therapies are emerging modalities that may enhance muscle flexibility, joint mobility, and neuromuscular activation, thereby contributing to athletic performance.

This randomized controlled study is designed to evaluate the effects of two different interventions-instrument-assisted soft tissue mobilization (IASTM) using the Graston technique, and percussion massage therapy using a handheld massage gun-on balance, explosive strength, and functional performance in competitive adolescent rowers aged 13-18. A total of 45 athletes meeting inclusion criteria will be randomly assigned to one of three groups: Vibration Group (percussion therapy at 33Hz), Soft Tissue Mobilization Group (IASTM), and Control Group (no intervention). Both interventions will be applied to the quadriceps femoris and gastrocnemius muscles over standardized durations and protocols.

Functional outcomes will be measured using the Y Balance Test, vertical jump test, single-leg hop tests (single, triple, crossover, square hop), and a 6-meter timed hop. Muscle strength will be evaluated using a myometer to assess isometric force production of the quadriceps and gastrosoleus muscles. Assessments will be conducted pre- and post-intervention.

The study is expected to provide clinically relevant data on the efficacy of myofascial techniques in enhancing functional capacity and performance parameters in young elite athletes. Findings may support the incorporation of soft tissue techniques and vibration therapy into performance training and injury prevention protocols for rowing and similar sports.

ELIGIBILITY:
Inclusion Criteria:

* Age between 13 and 18 years
* Licensed rowing athlete for at least 2 years
* Participating in at least 4 training sessions per week
* No lower extremity injury in the past 6 months
* Voluntary participation and signed informed consent form

Exclusion Criteria:

* History of surgery in the knee, hip, or ankle
* Neurological, vestibular, or systemic balance disorders
* Use of medications that may affect physical performance
* Orthopedic conditions that prevent participation in performance tests

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2025-06-13 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Y Balance Test Composite Score | Pre-intervention and immediately post-intervention
  Assesses dynamic balance and postural control of the lower extremities. During the test, participants perform maximal reach in three directions-anterior, posteromedial, and posterolateral-while maintaining a single-leg stance. The composite score is calculated by averaging the reach distances in all three directions, normalized to the participant's leg length using the formula:
  Composite Score = (Anterior + Posteromedial + Posterolateral) / (3 × limb length) × 100 Scale Range: 0 to 100% Interpretation: Higher scores indicate better dynamic balance and greater postural control.

SECONDARY OUTCOMES:
Vertical Jump Height | Pre-intervention and immediately post-intervention
  Measures lower extremity explosive strength. Participants perform a countermovement jump, and the maximum vertical jump height is recorded.
  Unit of Measure: centimeters (cm) Scale Range: Not fixed (depends on physical capacity; typically 10-80 cm) Interpretation: Higher scores indicate greater explosive power in the lower extremities.
Single-Leg Hop Tests | Pre-intervention and immediately post-intervention
  Assesses unilateral functional lower limb performance and dynamic stability. Participants perform a maximal forward hop on one leg, and the distance is measured.
  Unit of Measure: centimeters (cm) Scale Range: Not fixed (typically 50-250 cm) Interpretation: Greater distances reflect better functional strength and neuromuscular control.
6-Meter Timed Hop Test | Pre-intervention and immediately post-intervention
  Assesses power, speed, and dynamic control over a short distance using a single-leg hop. Total time to complete 6 meters is recorded.
Isometric Muscle Strength of Quadriceps and Gastrocnemius | Pre-intervention and immediately post-intervention
  Assessed with a hand-held myometer to measure maximal isometric force in Newtons.Myometer device with standard positioning and stabilization.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Dansuk, PhD, Principal Investigator — Medipol University
Locations (1):
- Tayfun Arslan, Sinop, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Menek B, Dansuk E, Arslan T. The Effects of Soft Tissue Mobilization and Vibration Therapy on Balance, Explosive Strength, and Functional Performance in Elite Rowers. J Strength Cond Res. 2025 Dec 5. doi: 10.1519/JSC.0000000000005305. Online ahead of print. PMID 41369532